CLINICAL TRIAL: NCT00692653
Title: Personal Patient Profile Prostate (P4) Randomized, Multisite Trial
Acronym: P4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Donna Berry, PhD, RN, FAAN, ACON, Director, The Phyllis F. Cantor Center, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R01NR009692 (NIH); R01NR009692 (NIH)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: Localized prostate cancer; Treatment decision making; Tailored decision aid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P4 (Experimental): Participant uses P4 program before meeting with his clinician to discuss treatment options.
  Interventions: Behavioral: P4
- Usual care+ (No Intervention): Usual care plus participant is directed to reputable websites highly rated in research literature to learn more about prostate cancer treatments.

INTERVENTIONS:
Behavioral: P4 — Tailored online decision support system for prostate cancer treatment decision making
  Arms: P4

SUMMARY:
The purpose of this study is to determine whether or not participation in an experimental program called the "P4 program" is useful to men who are faced with choices about treatment for their early stage prostate cancer. The P4 program consists of a series of questions and information for the participant.

Before seeing the cancer specialist, participants will answer several questionnaires on a computer. This will take about 20-30 minutes. Participants may choose to do this on a computer at home or on a touch-screen computer in the clinic. Half the participants will then be shown several highly rated informational websites about prostate cancer treatments. The other half, based on the individual participant's answers, will receive the P4 program's customized written and on-screen information. Reading the information and watching videos will take about 20 minutes.

About one month later, and again 6 months, participants will complete follow-up questionnaires electronically or by mail. These questionnaires will help us understand how each participant's decision for treatment of their prostate cancer went. Answering these questionnaires should take about 20 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of prostate cancer, stage I or II
* Diagnosis within the past 6 months
* Has appointment with a consulting specialist at one of the clinical trial sites
* Must be able to read and write English or Spanish at a 6th grade level
* Must not have begun any treatment (except watchful waiting)
* Must be able to complete baseline assessment before target clinician visit.

Exclusion Criteria:

* Advanced prostate cancer
* Diagnosed more than 6 months ago
* Cannot read and write English or Spanish at a 6th grade level
* Does not have appointment at one of the clinical trial sites

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict | Baseline to 6 months
Decisional Satisfaction | Baseline to 6 months
Satisfaction with Preparation for Decision Making | Baseline to 1 month

SECONDARY OUTCOMES:
Shift in decisional control preference from pre-decision to 1 month post-treatment | Baseline to 1 month
Resource utilization | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth Wolpin, RN, PhD, Principal Investigator — University of Washington; Donna L Berry, RN, PhD, Study Director — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - VA Medical Center / Medical College of Georgia, Augusta, Georgia
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Seattle Prostate Institute, Seattle, Washington
  - Veterans Administration Puget Sound Health Care System, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Underhill ML, Hong F, Berry DL. When study site contributes to outcomes in a multi-center randomized trial: a secondary analysis of decisional conflict in men with localized prostate cancer. Health Qual Life Outcomes. 2014 Oct 25;12:159. doi: 10.1186/s12955-014-0159-3. PMID 25344101
- [Derived] Bosco JL, Halpenny B, Berry DL. Personal preferences and discordant prostate cancer treatment choice in an intervention trial of men newly diagnosed with localized prostate cancer. Health Qual Life Outcomes. 2012 Sep 28;10:123. doi: 10.1186/1477-7525-10-123. PMID 23021156
- [Derived] Berry DL, Wang Q, Halpenny B, Hong F. Decision preparation, satisfaction and regret in a multi-center sample of men with newly diagnosed localized prostate cancer. Patient Educ Couns. 2012 Aug;88(2):262-7. doi: 10.1016/j.pec.2012.04.002. Epub 2012 May 17. PMID 22608696